CLINICAL TRIAL: NCT03926325
Title: Baseline Investigation of Patients With Cardiac Arrest in China
Acronym: BASIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Hainan Medical College (Other); Jinan Emergency Medical Center (Unknown); Wenshang County People's Hospital (Unknown); The Affiliated Hospital of Xuzhou Medical University (Other); Xuzhou Ambulance Center (Unknown); The First Affiliated Hospital of Anhui Medical University (Other); Hefei Emergency Medical Center (Unknown); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Hangzhou Emergency Medical Center (Unknown); RenJi Hospital (Other); Shanghai Changzheng Hospital (Other); Shanghai Emergency Medical Center (Unknown); First Affiliated Hospital of Fujian Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); China-Japan Friendship Hospital (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Beijing Friendship Hospital Affiliated to the Capital University of Medical Sciences (Unknown); Beijing Children's Hospital (Other); Beijing Emergency Medical Center (Other); Beijing Red Cross Emergency Rescue Center (Unknown); Tianjin Medical University General Hospital (Other); Tianjin Emergency Medical Center (Unknown); The Affiliated Hospital of Inner Mongolia Medical University (Other); Hohhot 120 Emergency Medical Center (Unknown); Siziwang Banner People's Hospital of Inner Mongolia (Unknown); First Hospital of Qinhuangdao (Unknown); Qinhuangdao Emergency Dispatching Center (Unknown); The First Affiliated Hospital of Shanxi Medical University (Other); Taiyuan Emergency Medical Center (Unknown); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Guangzhou Emergency Medical Command Center (Unknown); Haikou Emergency Medical Center (Other); People's Hospital of Wanning (Unknown); First Affiliated Hospital of Guangxi Medical University (Other); Nanning Emergency Medical Center (Unknown); Renmin Hospital of Wuhan University (Other); Wuhan Emergency Medical Center (Unknown); Qianjiang Central Hospital (Unknown); Henan Provincial People's Hospital (Other); Zhenzhou Emergency Medical Center (Unknown); Hunan Provincial People's Hospital (Other); The First Hospital of Jilin University (Other); Changchun Emergency Medical Center (Unknown); Nong'an County People's Hospital (Unknown); First Hospital of China Medical University (Other); Shenyang Emergency Center (Unknown); First Affiliated Hospital of Harbin Medical University (Other); Heilongjiang Emergency Medical Center (Unknown); Santai County People's Hospital (Unknown); Chongqing Emergency Medical Center (Other); Emergency Center of Yunan Province (Unknown); The Affiliated Hospital Of Guizhou Medical University (Other); Nyingchi People's Hospital (Unknown); First Affiliated Hospital of Xinjiang Medical University (Other); Lanzhou University Second Hospital (Other); Wushan County People's Hospital (Unknown); People's Hospital of Ningxia Hui Autonomous Region (Other); Yinchuan Emergency Medical Center (Unknown); Qinghai People's Hospital (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Xi'an Emergency Medical Center (Unknown); Fudan University (Other); National Center for Cardiovascular Disease (Unknown); Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other); Tiantan Hospital, Capital Medical University (Unknown); Peking University Third Hospital (Other); Beijing Chao Yang Hospital (Other); National Center for Chronic and Noncommunicable Disease Control and Prevention, China CDC (Other); National Health Commission of the People's Republic of China, Statistical information center (Unknown); Xiangya Hospital of Central South University (Other); West China Hospital (Other); Chang shu No.1 People's Hospital (Unknown)
Responsible Party: Principal Investigator, Feng Xu, Director of Emergency Department, Qilu Hospital of Shandong University
Other Study IDs: QLEmer201904
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — blood samples of cardiac arrest patients in certain centers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BASIC is a perspective, multicentre and large-scale registry focusing on of patients suffering a cardiac arrest in China. The aims of the study are to establish the monitoring sites covering out-of-hospital cardiac arrest (OHCA) and in-hospital cardiac arrest (IHCA) in urban and rural areas in 7 regions (East China, North China, South China, Central China, Northeast China, Southwest China and Northwest China) around China, to collect data from cardiac arrest patients, and to describe basic characteristics, treatments, outcomes, incidences and risk factors of OHCA and IHCA in China.

ELIGIBILITY:
Inclusion Criteria:

1. OHCA: Every patient who suffered a cardiac arrest that occurred in any location other than a hospital, and was attended and/or treated by an EMS.
2. IHCA: Every patient who suffered a cardiac arrest in hospital.
3. the representative population-based survey: Every patient who suffered a cardiac arrest in the selected cities or suburbs.

Exclusion Criteria:

1. OHCA: 1)The out-of-hospital cardiac arrest patients who were taken to the hospital by their family members; 2) Bystanders suspected cardiac arrest, but the ROSC was achieved without defibrillation or resuscitation by EMS.
2. IHCA: The patient who suffered a cardiac arrest that occurred out-of-hospital and then transferred to the hospital.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutive patients with cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of OHCA treated by EMS | Latest data inclusion June 30, 2022
incidence of IHCA | Latest data inclusion June 30, 2022
survival to hospital discharge or 30d survival of OHCA | at hospital discharge, 30days after cardiac arrest occurs
survival to hospital discharge or 30d survival of IHCA | at hospital discharge, 30days after cardiac arrest occurs
prevalence of favorable neurological outcome after cardiac arrest according to Cerebral Performance Category (CPC) Scale | at hospital discharge, 30days after cardiac arrest occurs
  CPC 1 and 2 as a favorable neurological outcome; CPC 1, Good Cerebral Performance; CPC 2, Moderate Cerebral Disability; CPC 3, Severe Cerebral Disability; CPC 4, Coma, vegetative state; CPC 5, Brain death

SECONDARY OUTCOMES:
survival of OHCA | 6 months and 1 year after cardiac arrest occurs
survival of IHCA | 6 months and 1 year after cardiac arrest occurs
prevalence of favorable neurological outcome after cardiac arrest according to Cerebral Performance Category (CPC) Scale | 6 months and 1 year after cardiac arrest occurs
  CPC 1 and 2 as a favorable neurological outcome; CPC 1, Good Cerebral Performance; CPC 2, Moderate Cerebral Disability; CPC 3, Severe Cerebral Disability; CPC 4, Coma, vegetative state; CPC 5, Brain death
rate of return of spontaneous circulation | Latest data inclusion June 30,2022

CONTACTS AND LOCATIONS:
Overall Officials: Feng Xu, Dr, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Xie X, Zheng J, Zheng W, Pan C, Ma Y, Zhu Y, Tan H, Han X, Yan S, Zhang G, Li C, Shao F, Wang C, Zhang J, Bian Y, Ma J, Cheng K, Liu R, Sang S, Zhang Y, McNally B, Ong MEH, Lv C, Chen Y, Xu F; BASIC-OHCA Coordinators and Investigators. Efforts to Improve Survival Outcomes of Out-of-Hospital Cardiac Arrest in China: BASIC-OHCA. Circ Cardiovasc Qual Outcomes. 2023 Feb;16(2):e008856. doi: 10.1161/CIRCOUTCOMES.121.008856. Epub 2022 Dec 12. PMID 36503279